CLINICAL TRIAL: NCT00389415
Title: A Multicenter, Open, Long Term Safety Study of 52 Weeks Treatment With Vildagliptin (100 mg qd) In Patients With Type 2 Diabetes (Extension Study of Study CLAF237A1303)
Brief Title: Long Term Safety of Vildagliptin (100mg qd) In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A1303E1
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Vildagliptin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This 52-week multicenter open-labeled extension study is designed to assess the long-term safety of vildagliptin (100 mg qd) in patients with Type 2 Diabetes. This extension study is open to patients who have completed core study CLAF237A1303.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as Type 2 Diabetes
* Patients who have completed study CLAF237A1303
* Outpatients

Exclusion Criteria:

* Patients who prematurely discontinued Study CLAF237A1303
* Other protocol-defined inclusion/exclusioncriterial may apply

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-10

PRIMARY OUTCOMES:
Adverse events profile after 52 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline to endpoint on HbA1c at 52 weeks
Change from baseline to endpoint on fasting plasma glucose at 52 weeks
Change from baseline to endpoint in HOMA B at 52 weeks
Change from baseline to endpoint in HOMA IR at 52 weeks
Change from baseline to endpoint in body weight at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan